CLINICAL TRIAL: NCT03384576
Title: The Effect of Music in the Pediatric Emergency Department Waiting Room on Caregiver Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jennifer Smedley, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 300001035
Record Dates: First submitted 2017-12-08; First posted 2017-12-27 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Anxiety
Keywords: Music; Emergency; caregivers
MeSH Terms: conditions — Anxiety Disorders; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music intervention (Experimental): Participants listen to music in the waiting room
  Interventions: Other: Music intervention
- No music (Active Comparator): Participants will not have music in the waiting room
  Interventions: Other: No music

INTERVENTIONS:
Other: Music intervention — Classical music to be played in the Emergency waiting room
  Arms: Music intervention
Other: No music — No music played in emergency waiting room
  Arms: No music

SUMMARY:
The purpose of this research study is to examine the effects of playing classical music in the waiting room on caregiver anxiety. People who enter the study will be asked a few identifier questions including age and relation to patient and then will be asked fill out a survey regarding anxiety.

DETAILED DESCRIPTION:
The study investigators will initially screen for participants based on the patient's acuity level. If the patient meets the low acuity requirement and if they have a wait time greater than 20 minutes then the caregiver will be approached to obtain informed consent once they have been placed in a room. If they choose to be included in the study, the patient's medical record number will be recorded, a personal identification number will be assigned, and the patient's information will be entered into the personal identification number key and into our research database. A questionnaire asking participants age and relation to patient and the state-trait anxiety inventory will be administered to the caregiver. An additional question of perceived wait time will also be asked.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers; age >18 year, accompanying a pediatric patient with acuity level ≥ 4
* Patient must have been in waiting area for at least 20 minutes

Exclusion Criteria:

* Non-english speaking caregivers
* Hearing impaired caregivers
* Caregivers accompanying a patient with an acuity level less than 4

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
reduction in anxiety score | up to 10 hours
  Participants will be administered with the State Trait Anxiety Inventory questionnaire , Scores range from 20-80 with higher score indicates greater anxiety

SECONDARY OUTCOMES:
Perceived waiting time | up to 10 hours
  Participants will be asked about perceived waiting time

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Smedley, DO, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No